CLINICAL TRIAL: NCT00502385
Title: Phase I AZD2171 in Patients With Relapsed or Refractory AML and Elderly Patients With DeNovo or Secondary AML
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D8480C00002
Record Dates: First submitted 2007-07-13; First posted 2007-07-17 (Estimated); Last update posted 2011-01-21 (Estimated); Status verified 2011-01

CONDITIONS: Leukaemia; Myelocytic; Acute
Keywords: Phase I; AML; de novo or secondary AML; AZD2171
MeSH Terms: conditions — Leukemia | interventions — cediranib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: AZD2171

SUMMARY:
The study will be conducted across multiple European centres to assess the safety and tolerability of multiple doses of AZD2171 in patients with AML.

ELIGIBILITY:
Inclusion Criteria:

* Provision of written informed consent
* Male/female, 18 yrs or over
* WHO performance status 0-2
* Disease not responding to or relapsing after chemotherapy or elderly patients not suited to chemotherapy

Exclusion Criteria:

* Acute myeloid leukaemia arising from previous chronic myeloid leukaemia or acute myeloid leukaemia of type FAB M3
* Previous treatment against new blood vessel formation (anti-angiogenic)
* Chest X-ray showing leukaemia in the lungs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2004-04

PRIMARY OUTCOMES:
The primary objective is to determine the safety and tolerability of multiple oral doses of AZD2171 in AML patients by assessment of AEs, BP&pulse, heart rate respiration rate, EKG, clinical chemistry

SECONDARY OUTCOMES:
Efficacy, PK

CONTACTS AND LOCATIONS:
Overall Officials: Nick Botwood, BSc, MBBS, MRCP, MFPM, Study Director — AstraZeneca; Dieter Hoelzer, MD, PhD, Principal Investigator — Frankfurt University Hospital